CLINICAL TRIAL: NCT03402035
Title: Shock, Whole Blood and Assessment of TBI- S.W.A.T.- Linking Investigations in Trauma and Emergency Services (LITES) Task Order 2
Brief Title: Shock, Whole Blood, and Assessment of TBI S.W.A.T. (LITES TO 2)
Acronym: SWAT
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Sperry, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO17090104
Record Dates: First submitted 2017-12-14; First posted 2018-01-17 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-06

CONDITIONS: Hemorrhagic Shock; Traumatic Brain Injury
Keywords: Whole Blood Resuscitation
MeSH Terms: conditions — Shock, Hemorrhagic; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mechanistic Banked Samples Mechanistic Biomarkers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Whole Blood: Subjects at enrolling centers that utilize whole blood for hemorrhagic shock
- Component Therapy: Subjects at enrolling centers that utilize component therapy for hemorrhagic shock

SUMMARY:
The LITES Network is an operational trauma center consortium which has the expertise, track record and confirmed capabilities to conduct prospective, multicenter, injury care and outcomes research of relevance to the Department of Defense (DoD).

Hemorrhage and Traumatic Brain Injury (TBI) are responsible for the largest proportion of all trauma-related deaths. It is the poly-trauma patient who suffers both hemorrhagic shock and traumatic brain injury where a paucity of evidence exists to direct treatment, limiting the development of beneficial trauma practice guidelines.

The use of Whole Blood (WB) for early trauma resuscitation has been touted as the 'essential next step' in the evolution of trauma resuscitation. Despite its historical and more recent use, little is known regarding WB's benefit relative to the 'current practice' ratio-based blood component therapy in the acutely bleeding patient, and even less is known regarding its effects in patients with TBI.

AIM#1: Evaluate patient centered outcomes associated with early whole blood resuscitation practice as compared to component resuscitation in poly-trauma patients with hemorrhagic shock and further characterize outcome benefits in those with traumatic brain injury.

AIM#2: Characterize blood pressure and resuscitation endpoints during the acute resuscitation phase of care and the associated/attributable outcomes for traumatic brain injury in patients with hemorrhagic shock.

General Hypothesis #1: Whole blood resuscitation will be associated with improved mortality and resuscitation outcomes in poly-trauma patients and long term neurological outcome in those patients with traumatic brain injury as compared to those resuscitated with component therapy.

General Hypothesis #2: Differences in prehospital and acute phase resuscitation systolic blood pressure will be associated with differential outcomes in patients with traumatic brain injury at discharge and at 6 months.

Study Design: The LITES network will perform a multicenter, prospective, observational cohort study over a 4 year period to determine the impact of whole blood resuscitation in trauma patients with hemorrhagic shock at risk of large volume resuscitation with and without TBI. Early whole blood resuscitation will be compared to standard component resuscitation. The study will also further characterize blood pressure and resuscitation endpoints in poly-trauma patients with traumatic brain injury. Six Trauma sites with appropriate characteristics will be selected from 12 LITES Network sites across the country.

Study Setting: The study will be performed utilizing busy level I trauma centers within the LITES Network located across the country, at sites where either whole blood has currently been incorporated into standard of care or where component blood transfusion is being utilized for patients in hemorrhagic shock at risk for large volume resuscitation.

Study Population: The study will focus on patients who suffer blunt or penetrating injury, transported to a SWAT participating LITES trauma center with evidence of hemorrhagic shock at risk of large volume blood resuscitation.

DETAILED DESCRIPTION:
Background

The LITES Network is an operational trauma center consortium which has the expertise, track record and confirmed capabilities to conduct prospective, multicenter, injury care and outcomes research of relevance to the Department of Defense (DoD). Clinical trials from the point of injury in the prehospital arena through the trauma bay and operating theatre, thru ICU and beyond discharge are feasible and critical to the overall goals of the network. Novel capabilities include prehospital point of care testing for shock severity and sequential coagulopathy measurements. The network and leadership have a track record of Exception From Informed Consent (EFIC) trials and expertise with those injury subtypes including traumatic brain injury, hemorrhagic shock and coagulopathy of trauma, poly-trauma and severe extremity trauma. In addition to the track record and proven capabilities, the LITES Network uses a central IRB and efficient methods to minimize time, resources, cost and regulatory burdens and improve recruitment, consent rates and ease of data acquisition to promote successful execution of those task orders provided to the network from the DoD.

Traumatic injury represents an incredible health care burden in the United States and worldwide.1 Hemorrhage and Traumatic Brain Injury (TBI) are responsible for the largest proportion of all trauma-related deaths. Despite advances in trauma resuscitation and brain injury management, few therapeutic interventions are available to reduce the downstream morbidity and mortality attributable to these injury patterns. It is the poly-trauma patient who suffers both hemorrhagic shock and traumatic brain injury where a paucity of evidence exists to direct treatment, limiting the development of beneficial trauma practice guidelines.

Ongoing traumatic blood loss is complicated by trauma induced coagulopathy which results in further unbridled hemorrhage and resultant shock and organ dysfunction. Secondary to increasing evidence and knowledge, in-hospital resuscitation of traumatic hemorrhage has changed over the past decade to reduce the coagulopathic response to ischemia and tissue injury. The underlying principle of current resuscitation practice focuses on preventing or reversing the effects of coagulopathy with the early use of a balanced component transfusion strategy (1:1:1 - plasma: packed red blood cells: platelets). This reconstituted strategy has also been coined 'whole blood-like' resuscitation despite being inferior from a compositional standpoint relative to Whole Blood (WB). The use of WB was historically the gold standard for treating hemorrhagic shock during World War I and II, prior to sweeping changes in blood banking practice. The use of WB for early trauma resuscitation is making a resurgence, primarily based upon the military experience and has been touted as the 'essential next step' in the evolution of trauma resuscitation. Despite its historical and more recent use, little is known regarding WB's benefit relative to the 'current practice' ratio based blood component therapy in the acutely injured patients and even less is known regarding its effects in patients with TBI.

Permissive hypotension has been thought to improve outcome in injured patients with hemorrhagic shock in the prehospital and acute resuscitation phase of treatment allowing for the ability to obtain surgical control of bleeding while minimizing ongoing hemorrhage. Despite this benefit for hemorrhagic shock patients, hypotension has been consistently shown to be associated with worse outcomes in patients with TBI. Interestingly, newer animal data suggests permissive hypotension may be beneficial in a swine TBI model.The majority of prior, high level TBI trials have excluded patients with concomitant hemorrhagic shock. Prospective evidence and long term TBI outcome data are lacking for these complex poly-trauma patients and the most appropriate blood pressure and most efficacious resuscitation target for patients with TBI and acute hemorrhage remain poorly characterized.

Hypothesis #1A: Whole blood resuscitation will be associated with a lower 4 hour mortality in poly-trauma patients as compared to those resuscitated with component therapy.

Hypothesis #1B: Whole blood resuscitation will be associated with a lower incidence of 12 hour and 24 hour mortality, a lower incidence of death from exsanguination, incidence of MOF, nosocomial infection, improved transfusion ratios, lower overall blood transfusion requirements and shorter time to hemostasis as compared to those resuscitated with component therapy.

Hypothesis #1C: Whole blood resuscitation will be associated with an improved Glasgow Outcome Score-Extended at 6 months post injury as compared to those resuscitated with component therapy in patients with traumatic brain injury.

Hypothesis #2A: A nadir prehospital and acute phase resuscitation systolic blood pressure greater than or equal to 120 mmHg will be associated with improved traumatic brain injury outcomes at discharge and at 6 months.

Hypothesis #2B: The magnitude of the dose depth curve of systolic blood pressure during the prehospital and acute phase resuscitation will be associated with neurological outcome differences at discharge and at 6 months following traumatic brain injury.

Research Design and Methods

Study Design: The LITES Network will perform a multicenter, prospective, observational cohort study over a 4 year period to determine the impact of whole blood resuscitation in trauma patients with hemorrhagic shock at risk of large volume resuscitation with and without TBI. Early whole blood resuscitation will be compared to standard component resuscitation. The study will also further characterize blood pressure and resuscitation endpoints in poly-trauma patients with traumatic brain injury. Six trauma sites with appropriate characteristics will be selected from 12 network sites across the country.

Study Setting: The study will be performed utilizing busy level I trauma centers from within the LITES Network located across the country, at sites where either whole blood has currently been incorporated into standard of care or where component blood transfusion is being utilized for patients in hemorrhagic shock at risk for large volume resuscitation. Due to the paucity of trauma centers who are currently utilizing whole blood for trauma patients as standard of care, the potential to incorporate sites outside of the current LITES Network may be required over time.

ELIGIBILITY:
Inclusion Criteria:

Patients with blunt or penetrating injury who meet the following criteria: 1, 2, and 3

1. Has 2 or more of any of the following:

   1. Hypotension (systolic blood pressure ≤ 90 mmHg) in the prehospital or emergency department setting,
   2. Penetrating mechanism,
   3. Positive FAST abdominal ultrasound,
   4. Heart Rate ≥ 120 in the prehospital or emergency department setting.

   AND
2. Taken to the Operating Room (laparotomy, thoracotomy or vascular exploration) or Interventional Radiology within 60 minutes of arrival.

   AND
3. Need of blood/blood component transfusion in prehospital setting, ED or OR within 60 minutes of arrival.

Exclusion Criteria:

1. Age ≤ 14
2. CPR > 5 consecutive minutes without ROSC
3. Penetrating brain injury with brain matter exposed
4. ED death

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will focus on patients who suffer blunt or penetrating injury, transported to a SWAT participating LITES trauma center with evidence of hemorrhagic shock at risk of large volume resuscitation.
Sampling Method: Non-Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Whole Blood: Subjects that received whole blood for hemorrhagic shock
- Component Therapy: Subjects that received component therapy for hemorrhagic shock
Period: Overall Study
Arm/Group | Whole Blood | Component Therapy
Started | 624 | 427
Completed | 624 | 427
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole Blood | Component Therapy | Total
Number analyzed (Participants) | 624 | 427 | 1051
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35.0 [26.0 to 51.0] | 35.0 [25.0 to 47.0] | 35.0 [26.0 to 49.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 130 | 208
  Male | 546 | 297 | 843
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 225 | 139 | 364
  White | 280 | 235 | 515
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 119 | 53 | 172
Region of Enrollment [Number; unit: participants]
  United States | 624 | 427 | 1051

OUTCOME MEASURES:

1. Primary Outcome: 4 Hour Mortality
Description: mortality at 4 hours
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Blood | Component Therapy
Number analyzed (Participants) | 624 | 427
Participants | 50 | 32

2. Secondary Outcome: 24 Hour Mortality
Description: mortality at 24 hours
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Blood | Component Therapy
Number analyzed (Participants) | 624 | 427
Participants | 82 | 49

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Whole Blood | Component Therapy
All-Cause Mortality (participants affected / at risk) | 110/624 | 66/427
Serious Adverse Events (participants affected / at risk) | 87/624 | 48/427
Other Adverse Events (participants affected / at risk) | 0/624 | 0/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole Blood (N=624) | Component Therapy (N=427)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 49 (49) | 22 (22)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 38 (38) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT03402035/Prot_SAP_000.pdf